CLINICAL TRIAL: NCT00491127
Title: Phase II Study of Cisplatin With Gemcitabine in Fixed Dose Rate Infusion and Dexamethasone in Second-Line in Patients With Aggressive Non-Hodgkin's Lymphoma
Brief Title: Cisplatin With Gemcitabine With Dexamethasone in Patients With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6899; B9E-XM-S315
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Gemcitabine; Cisplatin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin
Drug: dexamethasone

SUMMARY:
The purpose of this study it to evaluate efficacy of gemcitabine with cisplatin and dexamethasone in patients with aggressive non-Hodgkin's lymphoma who have previously progressed on first line of chemotherapy with anthracyclines.

ELIGIBILITY:
Inclusion Criteria:

* The patients must have a histological diagnosis of aggressive non-Hodgkin's lymphoma including the following sub-categories of the WHO classification:

  * Diffuse large B-cell lymphoma and its variants (immunoblastic, Burkitt-like, sclerosis of mediastinum, large B-cell MALT, rich in T-cells and anaplastic B-cell lymphoma)
  * Peripheral T-cell lymphoma
  * Anaplastic lymphoma of large T-cells /null cells
* Patients are eligible if they have documented evidence of progression after prior first-line chemotherapy containing anthracyclines associated or not with Rituximab. Patients with refractory disease to first line of treatment are also eligible.
* ECOG PS (performance status) less than or equal to 2
* Presence of bidimensionally measurable disease in accordance with WHO criteria.

Exclusion Criteria:

* Involvement of the CNS.
* Any medical condition which contraindicates the degree of hydration required for the safe use of cisplatin.
* Intermediate degree lymphoma derived from the malignant transformation of a previous low-grade lymphoma.
* Active infection (in the opinion of the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-04; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To evaluate response rate

SECONDARY OUTCOMES:
To assess toxicity
Overall survival
Event-free survival
Progression - free survival
Disease - free survival
Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid, Spain

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com